CLINICAL TRIAL: NCT05449535
Title: Phase Ia Study to Evaluate the Tolerability, Safety, Pharmacokinetics, Preliminary Pharmacodynamics, and Immunogenicity of Single-dose JYB1904 in Healthy Chinese Subjects
Brief Title: Study of JYB1904 (an Anti-immunoglobulin E Antibody) in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JY20210115-Ia; CTR20220973 (Registry Identifier: National Medical Products Administration of China)
Record Dates: First submitted 2022-06-29; First posted 2022-07-08 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: JYB1904/JYB1904 Placebo Arm: dose escalation. Omalizumab Arm: one dose level .
Who Masked: Participant, Investigator
Masking Description: JYB1904/JYB1904 Placebo Arm: double-blind (participant and investigator); Omalizumab Arm: non-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JYB1904/JYB1904 Placebo (Experimental): single-dose; subcutaneous injection in the deltoid region of the upper arm.
  Interventions: Drug: JYB1904; Drug: JYB1904 Placebo
- Omalizumab (Active Comparator): single-dose; subcutaneous injection in the deltoid region of the upper arm.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: JYB1904 — Dosage form: injection, solution； Usage and dosage matching:dose 1, dose 2, dose 3, dose 4, dose 5; single-dose; subcutaneous injection in the deltoid region of the upper arm.
  Arms: JYB1904/JYB1904 Placebo
Drug: Omalizumab — Dosage form: injection, powder, lyophilized, for solution； Usage and dosage matching:dose 1; single-dose; subcutaneous injection in the deltoid region of the upper arm.
  Other Names: Xolair
  Arms: Omalizumab
Drug: JYB1904 Placebo — Dosage form: injection, solution； Usage and dosage matching:dose 1, dose 2, dose 3, dose 4, dose 5; single-dose; subcutaneous injection in the deltoid region of the upper arm.
  Arms: JYB1904/JYB1904 Placebo

SUMMARY:
This phase Ia study is meant to evaluate the tolerability, safety, pharmacokinetics, preliminary pharmacodynamics, and immunogenicity of single-dose JYB1904, an anti-immunoglobulin E (IgE) antibody, in healthy Chinese subjects.

DETAILED DESCRIPTION:
This first-in-human study with a dose-escalation design is meant to evaluate the tolerability, safety, pharmacokinetics, preliminary pharmacodynamics, and immunogenicity of single-dose JYB1904 in healthy Chinese subjects.

The sequential dose levels (sample size) of JYB1904 are set at five different dose, with additional two JYB1904 placebo subjects in each group. The active comparator is omalizumab (Xolair).

Dosage and administration: single-dose; subcutaneous injection in the deltoid region of the upper arm.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study and provide written informed consent voluntarily, and comply with the requirements;
2. Healthy Chinese subjects aged 18-50 years, male or female;
3. Normal or abnormal but without clinical significance reports of physical examinations, vital signs, clinical laboratory tests and others.

Exclusion Criteria:

1. Surgery history within 6 months prior to screening or any surgery schedule during the study;
2. Last visit in previous drug clinical trial within 3 months prior to screening;
3. Acute diseases occur or receive any medication during the screening period;
4. Other conditions unsuitable for the study confirmed by the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Baseline through 168 days post-dose
  Incidence and features of AEs assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Serum concentrations of JYB1904 and Omalizumab | Baseline through 168 days post-dose
  Serum JYB1904 and Omalizumab assessed by pre-specified methods, and related pharmacokinetic parameters analysis
Serum concentrations of total/free IgE | Baseline through 168 days post-dose
  Serum total/free IgE assessed by a pre-specified method, and related pharmacodynamic parameters analysis
Serum concentrations of anti-drug antibody (ADA) and neutralizing antibody (Nab) | Baseline through 168 days post-dose
  Serum ADA and Nab assessed by pre-specified methods, and related immunogenic features analysis

CONTACTS AND LOCATIONS:
Overall Officials: Guiling Chen, MD, Principal Investigator — Shulan (Hangzhou) Hospital
Locations (1):
- Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No